CLINICAL TRIAL: NCT00401258
Title: An Open-Label Trial of Duloxetine for the Treatment of Irritable Bowel Syndrome Without Comorbid Major Depressive Disorder
Brief Title: An Open-Label Trial of Duloxetine for the Treatment of Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Associate Director of Translational Neuroscience Research, Mclean Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-001723
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Results first posted 2010-08-27 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; irritable bowel syndrome; irritable bowel
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): 12-week, open-label trial of duloxetine in subjects with IBS.
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — 30mg oral duloxetine per day for one week, titrated up to 60mg per day at day 8, concluded by a one week taper period of 4 days of 30mg pills at the conclusion of the study, followed by 3 days on no medication (4+3 days=1 week), concluded with a post-taper follow-up appointment with a study physician.
  Other Names: Cymbalta

SUMMARY:
We hypothesize that duloxetine treatment will be associated with improvement in symptoms of IBS, particularly abdominal pain, in individuals without comorbid major depressive disorder.

During this 12-week, open-label, outpatient study, male and female subjects between the ages of 18 and 65 years who have been diagnosed with irritable bowel syndrome (IBS) will be treated with open-label duloxetine.

DETAILED DESCRIPTION:
IBS is a chronic gastrointestinal disorder characterized by abdominal pain, altered bowel habits, and abdominal bloating for which no organic cause can be determined. Duloxetine has demonstrated efficacy in the treatment of depression as well as in several pain syndromes including diabetic peripheral neuropathy and fibromyalgia. We hypothesize that it will be a safe and efficacious treatment for the symptoms of IBS, in particular abdominal pain.

We plan to study 15 male and female subjects between the ages of 18 and 65 years who have had gastrointestinal symptoms at least 2 days/week for greater than six months and who have been diagnosed with IBS by a physician. During the 12-week study, subjects will receive open-label duloxetine titrated up to 60mg/day. Subjects will be asked to complete a total of ten study visits during the 12-week study period. All study visits will be conducted at McLean Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Subjects must have been diagnosed with irritable bowel syndrome by a physician
* Subjects must have had gastrointestinal symptoms for 2 or more days per week for > 6 months

Exclusion Criteria:

* Lifetime history of bipolar disorder, psychotic disorder, or obsessive-compulsive disorder
* Current (within past 6 months) diagnosis of major depressive disorder or substance abuse disorder
* Active suicidal/homicidal ideation
* Pregnant women or women of child-bearing potential not using an approved methods of contraception
* Individuals with an unstable medical condition that in the opinion of the investigator would interfere with the interpretation of symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Brennan BP, Fogarty KV, Roberts JL, Reynolds KA, Pope HG Jr, Hudson JI. Duloxetine in the treatment of irritable bowel syndrome: an open-label pilot study. Hum Psychopharmacol. 2009 Jul;24(5):423-8. doi: 10.1002/hup.1038. PMID 19548294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements
Groups:
- Duloxetine, 60 mg Daily: Open-label duloxetine was administered for a duration of 12 weeks. Subjects received duloxetine 30 mg daily for 1 week followed by duloxetine 60 mg daily for 11 weeks.
Period: Overall Study
Arm/Group | Duloxetine, 60 mg Daily
Started | 15
Completed | 8
Not Completed | 7
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Pain, as Determined by Daily Pain Diaries (Patterned After Item 3 From the Brief Pain Inventory; Cleeland and Ryan, 1994).
Description: Subjects rated abdominal pain daily on a scale of 0-10 (0 being no pain and 10 being worst pain). The pain score at each visit represented the mean score from all days since the previous visit.
Time Frame: baseline and week 12
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
Units on a scale | -1.5 [-2.3 to -0.7]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Brief Pain Inventory
Description: The Brief Pain Inventory is a self-administered questionnaire used to evaluate the severity of a patient's pain and its interference with their life.
  Four items measure pain severity on a scale of 0-10, with 0 being absence of pain and 10 being severe pain. Seven items measure pain interference on a scale of 0-10, with 0 being absence of interference and 10 being severe interference.
  The sub scale of both sub scores ranges 0-40, with 0 indicating no pain/interference and 40 indicating severe pain/interference.
  The primary analysis for this outcome was assessed at each visit with a longitudinal repeated-measures random regression analysis assessing the rate of change of the measure during the treatment period. The model for the mean included a term for time (modeled as a continuous variable) and the measure effect was the estimated change in the outcome at week 12.
Time Frame: At each visit
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale
  Average pain severity | -1.5 [-2.3 to -0.7]
  Average pain interference | -1.6 [-2.1 to -1.1]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Average pain severity statistical analysis; Test type: Superiority or Other; p < .001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Duloxetine, 60 mg Daily; Average pain interference statistical analysis; Test type: Superiority or Other; p < .001, Mixed Models Analysis

3. Secondary Outcome: Short Form McGill Pain Questionnaire
Description: The Short Form McGill Pain Questionnaire is a self-administered questionnaire that measures pain intensity experienced by the patient. Scores on 15 descriptors are rated on an intensity scale of 0-3 (with 0 being no pain to 3 being severe pain), and has an overall score of between 0-45, with 0 being no pain and 45 being worst possible pain.
  The primary analysis for this outcome was assessed at each visit with a longitudinal repeated-measures random regression analysis assessing the rate of change of the measure during the treatment period. The model for the mean included a term for time (modeled as a continuous variable) and the measure effect was the estimated change in the outcome at week 12.
Time Frame: At each visit
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale | -2.37 [-4.27 to -0.47]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p = .001, Mixed Models Analysis

4. Secondary Outcome: Clinical Global Impression Scale
Description: The Clinical Global Impression Scale is a clinician-rated scale that evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  The primary analysis for this outcome was assessed at each visit with a longitudinal repeated-measures random regression analysis assessing the rate of change of the measure during the treatment period. The model for the mean included a term for time (modeled as a continuous variable) and the measure effect was the estimated change in the outcome at week 12.
Time Frame: At each visit
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale | -1.7 [-2.3 to -1.1]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

5. Secondary Outcome: Hamilton Depression Rating Scale
Description: The Hamilton Depression Rating Scale is a clinician-rated scale consisting of 17 questions designed to assess depressive symptoms. Scores of 0-7 are considered normal, 8-16 suggest mild depression, 17-23 moderate depression, and scores over 24 are indicative of severe depression. 52 is the maximum score.
Time Frame: At first visit only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale | 6.7 (2.2)

6. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale is a clinician-administered scale designed to assess the severity of symptoms of anxiety. There are 14 items, scored on a scale of 0 (not present) to 4 (severe). The total score range is 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe.
  The primary analysis of this scale was an endpoint analysis of the change from baseline.
Time Frame: At baseline and week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale | -3.3 [-6.3 to -0.4]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis

7. Secondary Outcome: Irritable Bowel Syndrome-Quality of Life Scale
Description: The Irritable Bowel Syndrome (IBS) Quality of Life Scale is a self-report quality of life measure specific to Irritable Bowel Syndrome that can be used to assess the impact of IBS and its treatment. There are 34 items summed and averaged for a total score between 0-100, with higher scores indicating better IBS specific quality of life.
  Each item measures one of eight sub scales - dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationships - and is rated on a scale of 1-5 indicating how much the subject agrees with the statement (1 is no agreement, 5 is extreme agreement).
  The primary analysis of this scale was an endpoint analysis of the change from baseline.
Time Frame: At baseline and week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale | 14.8 [8.9 to 20.8]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

8. Secondary Outcome: Sheehan Disability Scale
Description: The Sheehan Disability Scale is a brief, 5-item self-report tool that assess functional impairment in work/school, social life, and family life. Scores range from 0-10 in each subset, with 0 being unimpaired and 10 being highly impaired.
  The primary analysis of this scale was an endpoint analysis of the change from baseline.
Time Frame: At baseline and week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine, 60 mg Daily
Number analyzed (Participants) | 15
units on a scale
  Work/School | -2.5 [-4.1 to -1.0]
  Social | -1.8 [-4.0 to 0.3]
  Family | -2.2 [-3.6 to -0.8]
Statistical Analysis 1: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — Refers to work/school sub-scale
Statistical Analysis 2: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p = 0.087, Mixed Models Analysis — Refers to social sub scale
Statistical Analysis 3: Comparison: Duloxetine, 60 mg Daily; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — Refers to family sub scale

ADVERSE EVENTS:
Arm/Group | Duloxetine, 60 mg Daily
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine, 60 mg Daily (N=15)
nausea (Gastrointestinal disorders) | 9 (9)
insomnia (Nervous system disorders) | 7 (7)
sedation (Nervous system disorders) | 4 (4)
constipation (Gastrointestinal disorders) | 6 (6)
anorgasmia (Reproductive system and breast disorders) | 2 (2)
dizziness (Nervous system disorders) | 2 (2)
dry mouth (Skin and subcutaneous tissue disorders) | 2 (2)
night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
tremor (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No